CLINICAL TRIAL: NCT04202263
Title: Assessment of Suppression of Cutaneous Allergic Responses and Pruritis by Topical Minocycline
Acronym: GINA3
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: State University of New York - Downstate Medical Center (Other)
Responsible Party: Principal Investigator, Rauno Joks, MD, Chief Division of Allergy Immunology, State University of New York - Downstate Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1476585
Record Dates: First submitted 2019-11-04; First posted 2019-12-17 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Allergic Rhinitis; Asthma
MeSH Terms: conditions — Rhinitis, Allergic; Asthma | interventions — Minocycline

STUDY DESIGN:
Intervention Model Description: Each subject will simultaneously be tested for responses to placebo (0%), 1%, 2% and 3% minocycline cream responses to induced allergic skin inflammation.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo cream without minocycline
  Interventions: Drug: Placebos
- Minocycline Arm (Active Comparator): Minocycline cream (1%,2%,3%)
  Interventions: Drug: Minocycline Topical

INTERVENTIONS:
Drug: Minocycline Topical — Placement of minocycline cream 0%, 1%, 2% or 3% at one of four identical allergen skin test sites.
  Other Names: minocycline
  Arms: Minocycline Arm
Drug: Placebos — Placement of minocycline cream 0%
  Other Names: Minocycline 0%
  Arms: Placebo

SUMMARY:
Adults with known respiratory allergy/asthma with known skin test sensitization will undergo repeat skin prick testing at 4 areas of both arms (bilateral forearms, bilateral upper arms). Each site will be challenged with up to three known allergens, saline and histamine controls. Mean wheal diameter after 20 minutes challenge will be determined. This is followed by placement of minocycline cream (0%, 1%, 2%, 3%), placed in randomized fashion at each of 1 of 4 skin test sites. Measurement of subsequent wheal diameter will be done at 30 minutes, 60 minutes and 24 hours.

DETAILED DESCRIPTION:
Adults with known respiratory allergy/asthma with known skin test sensitization will undergo repeat skin prick testing at 4 areas of both arms (bilateral forearms, bilateral upper arms). Each site will be challenged with up to three known allergens, saline and histamine controls. Mean wheal diameter after 20 minutes challenge will be determined. This is followed by placement of minocycline cream (0%, 1%, 2%, 3%), placed in randomized fashion at each of 1 of 4 skin test sites. Measurement of subsequent wheal diameter will be done at 30 minutes, 60 minutes and 24 hours.

In addition, itch assessment at each site will be done at baseline, 30 minutes, 60 minutes and 24 hours using VAS and questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Adult ( ages 18-75) outpatients with diagnosis of allergic rhinoconjunctivitis and/or asthma who have previously undergone epicutaneous skin prick testing with detection of at least one allergen positive.

Exclusion Criteria:

* Subjects who are unable/unwilling to undergo cessation of oral antihistamines for five days prior to testing.
* Current use of oral steroids or other systemic immunosuppressants, including omalizumab (anti-IgE therapy) and anti-IL-5 therapy.
* Allergic asthmatics who have current uncontrolled asthma.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2019-09-26 (Actual); Primary Completion 2023-09-25 (Estimated); Study Completion 2023-09-25 (Estimated)

PRIMARY OUTCOMES:
Change in mean diameter of treatment induced effect on wheal size | 24 hours
  Compare mean diameter of placebo associated mean wheal diameter vs. 1%, 2%, and 3% minocycline cream

SECONDARY OUTCOMES:
Change in itch scores by minocycline 1%, 2%, and 3% vs. placebo | 24 hours.
  Changes in both visual analogue scale (0 to 100mm, with greater itch being with higher scores) and verbal itch scores (0 to 3, with 0 being no itch and 3 being severe itch) with 1%, 2%,and 3% cream vs, placebo over time.

CONTACTS AND LOCATIONS:
Overall Officials: Rauno O Joks, Principal Investigator — State University of New York - Downstate Medical Center
Locations (1):
- SUNY Downstate Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No